CLINICAL TRIAL: NCT00370617
Title: An Efficacy and Safety Study Comparing Pegylated-Interferon and Ribavirin Plus Metformin to Pegylated-Interferon and Ribavirin in the Treatment of naïve Patients With Genotype 1 Chronic HCV Infection and Insulin Resistance
Brief Title: Pegylated-Interferon and Ribavirin Plus Metformin in the Treatment of Chronic HCV Infection and Insulin Resistance
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: METVIRAL
Record Dates: First submitted 2006-08-30; First posted 2006-08-31 (Estimated); Last update posted 2006-11-14 (Estimated); Status verified 2006-11

CONDITIONS: Chronic Hepatitis C; Insulin Resistance
Keywords: chronic hepatitis C; insulin resistance; therapy
MeSH Terms: conditions — Hepatitis C, Chronic; Insulin Resistance | interventions — Metformin

INTERVENTIONS:
Drug: metformin

SUMMARY:
Chronic hepatitis C virus (HCV) infection is associated with an increased risk for the development of type 2 diabetes and HCV infection itself may promote insulin resistance, irrespective of the severity of liver disease.

Insulin resistance seems to be genotype specific and may play a role in fibrogenesis in chronic hepatitis C.

In an "in vitro" model, increased levels of insulin may promote increased HCV replication.

RATIONALE Decreased insulin resistance and reduced hyperinsulinemia may facilitate the efficacy of anti-viral drugs on HCV replication.

DETAILED DESCRIPTION:
Chronic hepatitis C virus (HCV) infection is associated with an increased risk for the development of type 2 diabetes and HCV infection itself may promote insulin resistance, irrespective of the severity of liver disease.

* In patients with HCV infection, an increase in fasting insulin levels is associated with the presence of serum HCV core, the severity of hepatic fibrosis and a decrease in expression of insulin receptor substrate (IRS) 1 and IRS2, central molecules of the insulin-signaling cascade. Down-regulation of IRS1 and IRS2 has also been observed in HCV core-transgenic mice livers and HCV core-transfected human hepatoma cells.
* High levels of tumor necrosis factor-alpha, which acts by disturbing tyrosine phosphorylation of insulin receptor substrate-1, may be associated with insulin resistance both in animal models and in HCV patients.

Insulin resistance seems to be genotype specific and may play a role in fibrogenesis in chronic hepatitis C.

* In patients infected with genotype non-3, insulin resistance is associated with the degree of fibrosis, the rate of fibrosis progression and previous failed antiviral treatment.
* Insulin resistance, fibrosis, and genotype are independent predictors of the response to antiviral therapy in chronic hepatitis C patients treated with peginterferon plus ribavirin. A sustained virological response is achieved in 33% of patients with genotype 1 and insulin resistance compared with 60% of genotype 1 patients without insulin resistance.
* Insulin resistance is associated with a 3-fold risk of failure to antiviral treatment in patients with genotype 1 In an "in vitro" model, increased levels of insulin may promote increased HCV replication.

RATIONALE Decreased insulin resistance and reduced hyperinsulinemia may facilitate the efficacy of anti-viral drugs on HCV replication.

INDICATION Genotype 1 Chronic HCV hepatitis (CHC) associated with insulin resistance (IR).

OBJECTIVES To compare the efficacy and safety of Pegylated-Interferon and Ribavirin plus metformin to Pegylated-Interferon and Ribavirin for treatment of naïve patients with Genotype 1 Chronic HCV infection and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

1. No previous antiviral treatment
2. Persistently elevated alanine aminotransferase (ALT) and quantifiable HCV-RNA (>2000 copies/ml)
3. Liver biopsy (within 12 months) consistent with CHC with or without cirrhosis
4. Compensated liver disease (Child-Pugh grade A)
5. Insulin resistance (evaluated by HOMA-R and OGTT)
6. Negative pregnancy test

Exclusion Criteria:

1. Type 2 Diabetes (according to ADA criteria)
2. BMI > 30
3. Alcohol consumption > 30 g/day
4. Other forms of liver disease (HBV, autoimmune, genetic), HIV infection.
5. Anemia
6. Psychiatric disease
7. Thyroid disease poorly controlled
8. Overt cirrhosis, hepatocellular carcinoma
9. Significant cardiac, renal, pulmonary disease, seizures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2006-09; Study Completion 2009-01

PRIMARY OUTCOMES:
Combined end-point of non-detectable serum HCV-RNA (<100 copies/mL) and
normal serum ALT activity at the end of the 24 week treatment-free follow up period

SECONDARY OUTCOMES:
End-of-treatment virological and biochemical response
Sustained virological and biochemical response
End-of-treatment improvement of insulin resistance
End-of-treatment improvement of liver histology

CONTACTS AND LOCATIONS:
Overall Officials: Mario Rizzetto, MD, Principal Investigator — University of Torino
Locations (1):
- Division of Gastroenterology, University of Torino, Ospedale San Giovanni Battista, Torino, Italy

REFERENCES:
- [Background] Romero-Gomez M, Del Mar Viloria M, Andrade RJ, Salmeron J, Diago M, Fernandez-Rodriguez CM, Corpas R, Cruz M, Grande L, Vazquez L, Munoz-De-Rueda P, Lopez-Serrano P, Gila A, Gutierrez ML, Perez C, Ruiz-Extremera A, Suarez E, Castillo J. Insulin resistance impairs sustained response rate to peginterferon plus ribavirin in chronic hepatitis C patients. Gastroenterology. 2005 Mar;128(3):636-41. doi: 10.1053/j.gastro.2004.12.049. PMID 15765399